CLINICAL TRIAL: NCT00698958
Title: A Randomized Trial to Compare the Effectiveness of Hospital or Ambulatory Approach for Adaptation to Non-Invasive Mechanical Ventilation in Patients With Chronic Respiratory Failure Secondary to Neuromuscular Diseases or Thoracic Cage Alterations
Brief Title: Ambulatory Adaptation to Non-Invasive Mechanical Ventilation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: Hospital Universitari Vall d'Hebron Research Institute (Other); Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Xavier Muñoz Gall, Hospitals Vall d'Hebron
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NEUMO/2002/01
Record Dates: First submitted 2008-06-13; First posted 2008-06-17 (Estimated); Last update posted 2008-06-17 (Estimated); Status verified 2008-06

CONDITIONS: Chronic Respiratory Failure
Keywords: Respiratory insufficiency; Hypercapnic chronic respiratory failure secondary to neuromuscular diseases or alterations of thoracic cage
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Hospital based adaptation to non- invasive mechanical ventilation for 7 days
  Interventions: Procedure: Hospital based adaptation to non- invasive mechanical ventilation for 7 days
- 2 (Experimental): Ambulatory adaptation to non- invasive mechanical ventilation for 7 days
  Interventions: Procedure: Ambulatory adaptation to non- invasive mechanical ventilation for 7 days

INTERVENTIONS:
Procedure: Ambulatory adaptation to non- invasive mechanical ventilation for 7 days — Ambulatory adaptation to non- invasive mechanical ventilation for 7 days
  Arms: 2
Procedure: Hospital based adaptation to non- invasive mechanical ventilation for 7 days — Hospital based adaptation to non- invasive mechanical ventilation for 7 days
  Arms: 1

SUMMARY:
A randomised study to assess the effectiveness of ambulatory adaptation to non-invasive mechanical ventilation in patient with hypercapnic respiratory failure secondary to neuromuscular diseases or alterations in thoracic cage in comparison with hospital adaptation.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 75
2. Chronic respiratory insufficiency secondary to neuromuscular disease or thoracic cage alterations with indication of non-invasive mechanical ventilation (presence of fatigue, dyspnea, morning headache, etc) plus one of the following criteria):

   * PaCO2 > 45 mmHg
   * Night time oxygen saturation < 88% at least for 5 consecutive minutes
   * In neuromuscular diseases, PIM < 60 cmH2O or FVC < 50% of theoretical.
3. Stable disease.
4. Airway access through nasal mask.
5. Ability to provide written informed consent.
6. Ability to attend the visits

Exclusion Criteria:

1. Contraindications for mechanical ventilation:

   * Patient with terminal disease or vegetative state
   * Lack of motivation of the patient
   * Lack of family or social support
   * Patients clinically unstable
   * Agitation or lack of co-operation
   * Depression.
2. Patients with acute symptoms requiring hospital admission.
3. Need for airway access through tracheostomy, face mask or mouth piece.
4. Relevant comorbidity (ie. heart failure, diabetes non controlled, infections, malignancies, etc.) leading to difficulties in adaptation to ventilation.
5. Use (for 7 days or more) of CNS depressors(benzodiazepines, antihistamines H1, tricyclic antidepressants , antiepileptic or antipsychotic drugs ) in the 30-day period prior to inclusion, or expected need for such drugs during the study.
6. Lack of understanding of the study procedures.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2003-06

PRIMARY OUTCOMES:
Change in PaCO2 from baseline | 6 months

SECONDARY OUTCOMES:
Change in PaCO2 from start of mechanical ventilation
6-minute walking test
Adaptation failure

REFERENCES:
- [Derived] Pallero M, Puy C, Guell R, Pontes C, Marti S, Torres F, Anton A, Munoz X. Ambulatory adaptation to noninvasive ventilation in restrictive pulmonary disease: a randomized trial with cost assessment. Respir Med. 2014 Jul;108(7):1014-22. doi: 10.1016/j.rmed.2014.04.016. Epub 2014 May 2. PMID 24837977